CLINICAL TRIAL: NCT00402363
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Trial to Assess the Efficacy and Safety of Lovaza for the Prevention of Recurrent, Symptomatic Atrial Fibrillation
Brief Title: Evaluation of Efficacy and Safety of Lovaza (Omega-3-Acid Ethyl Esters) in Recurrent, Symptomatic Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OM8 Afib
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Fibrillation, Atrial
Keywords: Lovaza; Omega-3 fatty acids; Omacor; Paroxysmal atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega-3-acid ethyl esters (Experimental)
  Interventions: Drug: omega-3-acid ethyl esters
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: omega-3-acid ethyl esters
  Arms: omega-3-acid ethyl esters
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Omacor (omega-3-acid ethyl esters) in patients with recurrent, symptomatic atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or older
* History of symptomatic atrial fibrillation (either paroxysmal or persistent)
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Permanent (chronic) atrial fibrillation
* Antiarrhythmic drug therapy which cannot be stopped
* Use of amiodarone with prior 6 months
* History of unsuccessful cardioversion
* History of certain cardiovascular conditions or cardiac surgery within prior 6 months
* History of stroke within prior 6 months
* Implanted cardio-defibrillator
* Certain circulatory, thyroid, pulmonary, liver, kidney, musculoskeletal or metabolic conditions, or cancer (except non-melanoma skin cancer)
* Poorly controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (152):
- United States (152):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Cottonwood, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Alamada, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Merced, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Bridgeport, Connecticut
  - GSK Investigational Site, Farmington, Connecticut
  - GSK Investigational Site, Guilford, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Fort Meyers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hudson, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Bannockburn, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, La Porte, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Mount Sterling, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lacombe, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Biddeford, Maine
  - GSK Investigational Site, Portland, Maine
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Ayer, Massachusetts
  - GSK Investigational Site, Brookline, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Alpena, Michigan
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Mineappolis, Minnesota
  - GSK Investigational Site, Rochester Hills, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Kalispell, Montana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Wayne, New Jersey
  - GSK Investigational Site, Babylon, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Troy, New York
  - GSK Investigational Site, West Islip, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Grand Forks, North Dakota
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Bryan, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Fairview Park, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Corvalis, Oregon
  - GSK Investigational Site, Hillsboro, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Greensburg, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Langhorne, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Ridley Park, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Wynnewood, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Cranston, Rhode Island
  - GSK Investigational Site, Pawtucket, Rhode Island
  - GSK Investigational Site, Westerly, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Humble, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, Orange, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Galax, Virginia
  - GSK Investigational Site, Richlands, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Springfield, Virginia
  - GSK Investigational Site, Burien, Washington
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Beloit, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Kowey PR, Reiffel JA, Ellenbogen KA, Naccarelli GV, Pratt CM. Efficacy and safety of prescription omega-3 fatty acids for the prevention of recurrent symptomatic atrial fibrillation: a randomized controlled trial. JAMA. 2010 Dec 1;304(21):2363-72. doi: 10.1001/jama.2010.1735. Epub 2010 Nov 15. PMID 21078810
- [Derived] Pratt CM, Reiffel JA, Ellenbogen KA, Naccarelli GV, Kowey PR. Efficacy and safety of prescription omega-3-acid ethyl esters for the prevention of recurrent symptomatic atrial fibrillation: a prospective study. Am Heart J. 2009 Aug;158(2):163-169.e1-3. doi: 10.1016/j.ahj.2009.05.024. PMID 19619690
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: OM8 Afib — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxysmal AF, P-OM3: Participants with paroxysmal atrial fibrillation (AF) receiving P-OM3, 8 grams (g) per day for the first 7 days; 4 g per day thereafter through Week 24. Paroxysmal AF was defined as AF that had never been treated with pharmacologic/electrical therapy to terminate an episode. A documented episode of symptomatic paroxysmal AF was defined as AF documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF in the participant's medical record.
- Paroxysmal AF, Placebo: Participants with paroxysmal AF receiving matching placebo. Paroxysmal AF was defined as AF that had never been treated with pharmacologic/electrical therapy to terminate an episode. A documented episode of symptomatic paroxysmal AF was defined as AF documented by an ECG or TTM tracing associated with symptoms consistent with AF in the participant's medical record.
- Persistent AF, P-OM3: Participants with persistent AF receiving P-OM3, 8 g per day for the first 7 days; 4 g per day thereafter through Week 24. Persistent AF was defined as AF that had been terminated at least once with pharmacologic/electrical cardioversion. A documented episode of symptomatic persistent AF was defined as AF documented by an ECG or TTM tracing associated with symptoms consistent with AF in the participant's medical record.
- Persistent AF, Placebo: Participants with persistent AF receiving matching placebo. Persistent AF was defined as AF that had been terminated at least once with pharmacologic/electrical cardioversion. A documented episode of symptomatic persistent AF was defined as AF documented by an ECG or TTM tracing associated with symptoms consistent with AF in the participant's medical record.
Period: Overall Study
Arm/Group | Paroxysmal AF, P-OM3 | Paroxysmal AF, Placebo | Persistent AF, P-OM3 | Persistent AF, Placebo
Started | 266 | 276 | 66 | 55
Completed | 233 | 246 | 60 | 45
Not Completed | 33 | 30 | 6 | 10
Not completed — Adverse Event | 9 | 14 | 2 | 2
Not completed — Withdrew Consent | 10 | 5 | 2 | 1
Not completed — Protocol Violation | 3 | 5 | 0 | 3
Not completed — Lost to Follow-up | 5 | 4 | 0 | 2
Not completed — Captured as "Other" | 6 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxysmal AF, P-OM3 | Paroxysmal AF, Placebo | Persistent AF, P-OM3 | Persistent AF, Placebo | Total
Number analyzed (Participants) | 266 | 276 | 66 | 55 | 663
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (13.56) | 61.9 (11.57) | 58.7 (12.65) | 57.6 (14.85) | 60.5 (12.84)
Gender [Count of Participants; unit: Participants]
  Female | 119 | 138 | 14 | 19 | 290
  Male | 147 | 138 | 52 | 36 | 373
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 246 | 253 | 63 | 45 | 607
  African American | 10 | 10 | 2 | 6 | 28
  Hispanic | 9 | 9 | 1 | 3 | 22
  American Indian | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Unknown | 1 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Paroxysmal AF With an Event of Documented Symptomatic Atrial Fibrillation (AF)/Flutter
Description: A documented episode of symptomatic AF /Flutter was defined as AF/Flutter documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF. Atrial flutter, a closely related rhythm disorder, was distinguished from AF by the presence of distinctive flutter p-waves at regluar intervals. The occurrence of symptomatic atrial flutter was treated as an occurrence of symptomatic AF for this outcome measure. "Censored" in the table below refers to participants who did not have a documented episode of symptomatic AF or flutter.
Time Frame: From first dose of study drug (Day 1) to the first symptomatic recurrence of AF/flutter (up to Week 24)
Population: Modified Intent-to-Treat (MITT) Population: all randomized participants who provided at least one post-randomization TTM ECG data transfer or equivalent
Measure: Number; unit: participants
Groups:
- Paroxysmal AF, Placebo: Participants with paroxysmal AF receiving matching placebo
- Paroxysmal AF, P-OM3: Participants with paroxysmal atrial fibrillation (AF) receiving P-OM3, 8 g per day for the first 7 days; 4 g per day thereafter through Week 24
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3
Number analyzed (Participants) | 269 | 258
participants
  Participants with event | 129 | 135
  Censored participants | 140 | 123
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.263, Regression, Cox; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.90 to 1.46]

2. Secondary Outcome: Number of Participants With Persistent AF and in Both AF Subgroups Combined With an Event of Documented Symptomatic AF/Flutter
Description: A documented episode of symptomatic AF/flutter was defined as AF/flutter documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF. Atrial flutter, a closely related rhythm disorder, was distinguished from AF by the presence of distinctive flutter p-waves at regluar intervals. The occurrence of symptomatic atrial flutter was treated as an occurrence of symptomatic AF for this outcome measure. "Censored" in the table below refers to participants who did not have a documented episode of symptomatic AF or flutter.
Time Frame: From first dose of study drug (Day 1) to the first symptomatic recurrence of AF/flutter (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Groups:
- Persistent AF, Placebo: Participants with persistent AF receiving matching placebo
- Persistent AF, P-OM3: Participants with persistent atrial fibrillation (AF) receiving P-OM3, 8 g per day for the first 7 days; 4 g per day thereafter through Week 24
- Combined, Placebo: Participants with both paroxysmal and persistent AF receiving matching placebo
- Combined, P-OM3: Participants with both paroxysmal and persistent atrial fibrillation (AF) receiving P-OM3, 8 g per day for the first 7 days; 4 g per day thereafter through Week 24
Arm/Group | Persistent AF, Placebo | Persistent AF, P-OM3 | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 54 | 64 | 323 | 322
participants
  Participants with event | 18 | 32 | 147 | 167
  Censored participants | 36 | 32 | 176 | 155
Statistical Analysis 1: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.089, Log Rank; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.92 to 2.92]
Statistical Analysis 2: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.081, Regression, Cox; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.98 to 1.52]

3. Secondary Outcome: Number of Participants With Paroxysmal AF or Persistent AF With an Event of Documented Symptomatic AF (Exclusive of Atrial Flutter)
Description: A documented episode of symptomatic AF was defined as AF documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF. "Censored" in the table below refers to participants who did not have a documented episode of symptomatic AF.
Time Frame: From first dose of study drug (Day 1) to the first symptomatic recurrence of AF (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3
Number analyzed (Participants) | 269 | 258 | 54 | 64
participants
  Participants with event | 126 | 133 | 18 | 30
  Censored participants | 143 | 125 | 36 | 34
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.213, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.91 to 1.49]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.171, Log Rank; Hazard Ratio (HR) = 1.50, 95% CI 2-sided [0.83 to 2.69]

4. Secondary Outcome: Number of Participants in Both AF Subgroups Combined With an Event of Documented Symptomatic AF (Exclusive of Atrial Flutter)
Description: as for outcome 3
Time Frame: From first dose of study drug (Day 1) to the first symptomatic recurrence of AF (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Groups:
- Combined, Placebo: Participants with paroxysmal and persistent AF receiving matching placebo
- Combined, P-OM3: Participants with paroxysmal and persistent atrial fibrillation (AF) receiving P-OM3, 8 g per day for the first 7 days; 4 g per day thereafter through Week 24
Arm/Group | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 323 | 322
participants
  Participants with event | 144 | 163
  Censored participants | 179 | 159
Statistical Analysis 1: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.082, Regression, Cox; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.98 to 1.53]

5. Secondary Outcome: Number Participants With Paroxysmal or Persistent AF With an Event of Documented Symptomatic or Asymptomatic AF/Flutter
Description: A documented episode of symptomatic or asymptomatic AF/flutter was defined as AF/flutter documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF. Asymptomatic episodes of AF or flutter were recorded by TTM during routine bi-weekly transmissions. Atrial flutter, a closely related rhythm disorder, was distinguished from AF by the presence of distinctive flutter p-waves at regluar intervals. "Censored" in the table below refers to participants who did not have a documented episode of symptomatic or asymptomatic AF/flutter.
Time Frame: From first dose of study drug (Day 1) to the first symptomatic or asymptomatic recurrence of AF/flutter (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3
Number analyzed (Participants) | 269 | 258 | 54 | 64
participants
  Participants with event | 149 | 153 | 27 | 40
  Censored participants | 120 | 105 | 27 | 24
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.331, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.89 to 1.40]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.297, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.79 to 2.11]

6. Secondary Outcome: Number of Participants in Both AF Subgroups Combined With an Event of Documented Symptomatic or Asymptomatic AF/Flutter
Description: as for outcome 5
Time Frame: From first dose of study drug (Day 1) to the first symptomatic or asymptomatic recurrence of AF/flutter (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 323 | 322
participants
  Participants with event | 176 | 193
  Censored participants | 147 | 129
Statistical Analysis 1: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.168, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.94 to 1.42]

7. Secondary Outcome: Number of Participants With Paroxysmal or Persistent AF With an Event of Documented Symptomatic or Asymptomatic AF (Exclusive of Flutter)
Description: A documented episode of symptomatic or asymptomatic AF was defined as AF documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF. Asymptomatic episodes of AF were recorded by TTM during routine bi-weekly transmissions. "Censored" in the table below refers to participants who did not have a documented episode of symptomatic or asymptomatic AF/flutter.
Time Frame: From first dose of study drug (Day 1) to the first symptomatic or asymptomatic recurrence of AF (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3
Number analyzed (Participants) | 269 | 258 | 54 | 64
participants
  Participants with event | 146 | 151 | 27 | 38
  Censored participants | 123 | 107 | 27 | 26
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.270, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.90 to 1.43]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.486, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.73 to 1.95]

8. Secondary Outcome: Number of Participants in Both AF Subgroups Combined With an Event of Documented Symptomatic or Asymptomatic AF (Exclusive of Flutter)
Description: as for outcome 7
Time Frame: From first dose of study drug (Day 1) to the first symptomatic or asymptomatic recurrence of AF (up to Week 24)
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 323 | 322
participants
  Participants with event | 173 | 189
  Censored participants | 150 | 133
Statistical Analysis 1: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.167, Regression, Cox; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.94 to 1.42]

9. Secondary Outcome: Number of Participants With Paroxysmal or Persistent AF With an Event After Completion of Day 7 to the Occurrence of Symptomatic AF/Flutter
Description: A documented episode of symptomatic AF/flutter was defined as AF/flutter documented by an electrocardiogram (ECG) or transtelephonic monitoring (TTM) tracing associated with symptoms consistent with AF. Atrial flutter, a closely related rhythm disorder, was distinguished from AF by the presence of distinctive flutter p-waves at regluar intervals. "Censored" in the table below refers to participants who did not have a documented episode of symptomatic AF/flutter.
Time Frame: From completion of Day 7 of study drug to the first symptomatic recurrence of AF/flutter (up to Week 24)
Population: MITT Population. Participants with events that occurred in the first 7 days were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3
Number analyzed (Participants) | 224 | 205 | 49 | 57
participants
  Participants with event | 88 | 87 | 15 | 27
  Censored participants | 136 | 118 | 34 | 30
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.565, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.81 to 1.47]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.103, Log Rank; Hazard Ratio (HR) = 1.68, 95% CI 2-sided [0.89 to 3.15]

10. Secondary Outcome: Number of Participants in the Combined AF Subgroups With an Event After Completion of Day 7 to the Occurrence of Symptomatic AF/Flutter
Description: as for outcome 9
Time Frame: From completion of Day 7 of study drug to the first symptomatic recurrence of AF/flutter (up to Week 24)
Population: MITT Population. Participants with events that occurred in the first 7 days were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 273 | 262
participants
  Participants with event | 103 | 114
  Censored participants | 170 | 148
Statistical Analysis 1: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.185, Regression, Cox; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.92 to 1.56]

11. Secondary Outcome: Number of Participants With Paroxysmal or Persistent AF With an Event That Occurred After Completion of Day 7 to the Occurrence of Symptomatic AF (Exclusive of Flutter)
Description: as for outcome 3
Time Frame: From completion of Day 7 of study drug to the first symptomatic recurrence of AF (up to Week 24)
Population: MITT Population. Participants with events that occurred in the first 7 days were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3
Number analyzed (Participants) | 225 | 206 | 49 | 57
participants
  Participants with event | 86 | 86 | 15 | 25
  Censored participants | 139 | 120 | 34 | 32
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.461, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.83 to 1.51]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.206, Log Rank; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.79 to 2.86]

12. Secondary Outcome: Number of Participants in the Combined AF Subgroups With an Event That Occurred After Completion of Day 7 to the Occurrence of Symptomatic AF (Exclusive of Flutter)
Description: as for outcome 3
Time Frame: From completion of Day 7 of study drug to the first symptomatic recurrence of AF (up to Week 24)
Population: MITT Population. Participants with events that occurred in the first 7 days were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 274 | 263
participants
  Participants with event | 101 | 111
  Censored participants | 173 | 152
Statistical Analysis 1: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.188, Regression, Cox; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.92 to 1.57]

13. Secondary Outcome: Annualized Number of AF/Flutter Rescue Episodes During the Treatment Period
Description: Rescue was defined as any pharmacological/electrical/surgical intervention for the termination/prevention of AF/flutter with a maximum of one rescue episode counted per day. Note: all annualized values were calculated by counting the number of rescue episodes, dividing by the number of days on treatment, then multiplying that number by 365.25.
Time Frame: From first dose of study drug (Day 1) to the last dose of study drug (up to Week 24)
Population: MITT Population. The number analyzed represents those participants who had a rescue episode.
Measure: Median (Inter-Quartile Range); unit: rescue episodes
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3 | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 34 | 37 | 8 | 21 | 42 | 58
rescue episodes | 2.44 [2.15 to 4.40] | 4.17 [2.16 to 6.52] | 2.17 [2.12 to 3.16] | 2.24 [2.15 to 4.25] | 2.19 [2.12 to 4.35] | 4.01 [2.15 to 4.37]
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.290, non-parametric ANCOVA; median difference (Hodges-Lehmann) = 0.070, 95% CI 2-sided [-0.09 to 2.08]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.479, Wilcoxon (Mann-Whitney); median difference (Hodges-Lehmann) = 0.063, 95% CI 2-sided [-0.08 to 2.02]
Statistical Analysis 3: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.218, non-parametric ANCOVA; median difference (Hodges-Lehmann) = 0.039, 95% CI 2-sided [-0.06 to 1.49]

14. Secondary Outcome: Annualized Cumulative Frequency of Symptomatic AF/Flutter Recurrences During the Treatment Period
Description: Values were annualized by counting the number of episodes of symptomatic AF/flutter recurrences (maximum of one per day), dividing by the number of days on treatment, then multiplying this number by 365.25.
Time Frame: From first dose of study drug (Day 1) to the last dose of study drug (up to Week 24)
Population: MITT Population. The number analyzed represents those participants with an event.
Measure: Median (Inter-Quartile Range); unit: recurrences
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3 | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 129 | 140 | 19 | 34 | 148 | 174
recurrences | 6.81 [3.89 to 13.12] | 8.32 [4.17 to 16.80] | 4.22 [2.08 to 6.37] | 4.35 [2.19 to 10.62] | 6.48 [2.23 to 12.89] | 6.52 [3.93 to 15.22]
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.218, non-parametric ANCOVA; median difference (Hodges-Lehmann) = 0.321, 95% CI 2-sided [-0.18 to 2.21]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.188, Wilcoxon (Mann-Whitney); median difference (Hodges-Lehmann) = 0.216, 95% CI 2-sided [-0.14 to 3.14]
Statistical Analysis 3: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.097, non-parametric ANCOVA; median difference (Hodges-Lehmann) = 0.181, 95% CI 2-sided [-0.10 to 2.10]

15. Secondary Outcome: Annualized Cumulative Frequency of Symptomatic AF Recurrences During the Treatment Period
Description: Values were annualized by counting the number of episodes of symptomatic AF recurrences (maximum of one per day), dividing by the number of days on treatment, then multiplying this number by 365.25.
Time Frame: From first dose of study drug (Day 1) to the last dose of study drug (up to Week 24)
Population: MITT Population. The number analyzed represents those participants with an event.
Measure: Median (Inter-Quartile Range); unit: recurrences
Arm/Group | Paroxysmal AF, Placebo | Paroxysmal AF, P-OM3 | Persistent AF, Placebo | Persistent AF, P-OM3 | Combined, Placebo | Combined, P-OM3
Number analyzed (Participants) | 126 | 139 | 19 | 32 | 145 | 171
recurrences | 6.91 [2.23 to 13.12] | 8.30 [4.01 to 16.60] | 4.22 [2.08 to 6.37] | 4.35 [2.18 to 11.02] | 6.48 [2.17 to 12.89] | 6.52 [3.02 to 15.13]
Statistical Analysis 1: Comparison: Paroxysmal AF, Placebo vs Paroxysmal AF, P-OM3; Test type: Superiority or Other; p = 0.239, non-parametric ANCOVA; median difference (Hodges-Lehmann) = 0.242, 95% CI 2-sided [-0.19 to 2.17]
Statistical Analysis 2: Comparison: Persistent AF, Placebo vs Persistent AF, P-OM3; Test type: Superiority or Other; p = 0.152, Wilcoxon (Mann-Whitney); median difference (Hodges-Lehmann) = 0.249, 95% CI 2-sided [-0.09 to 4.31]
Statistical Analysis 3: Comparison: Combined, Placebo vs Combined, P-OM3; Test type: Superiority or Other; p = 0.094, non-parametric ANCOVA; median difference (Hodges-Lehmann) = 0.200, 95% CI 2-sided [-0.08 to 2.11]

ADVERSE EVENTS:
Time Frame: Day 1 through Week 24
Description: Serious adverse events (SAEs) and adverse events (AEs) were collected in the Safety Population, comprised of all participants who received and took at least one dose of study medication. Events reported are "treatment emergent," defined as an event of new onset or one that worsened during the on-treatment period.
Groups:
- Placebo: Participants receiving matching placebo
- Prescription Omega-3 Acid Ethyl Esters: Participants receiving P-OM3, 8 g per day for the first 7 days; 4 g per day thereafter through Week 24
Arm/Group | Placebo | Prescription Omega-3 Acid Ethyl Esters
Serious Adverse Events (participants affected / at risk) | 20/331 | 25/332
Other Adverse Events (participants affected / at risk) | 66/331 | 82/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=331) | Prescription Omega-3 Acid Ethyl Esters (N=332)
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal hematoma (Gastrointestinal disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
False positive tuberculosis test (Investigations) | 0 | 1
International normalized ratio increased (Investigations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 1 | 0
Suicide (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=331) | Prescription Omega-3 Acid Ethyl Esters (N=332)
Urinary tract infection (Infections and infestations) | 12 | 12
Sinusitis (Infections and infestations) | 12 | 10
Nasopharyngitis (Infections and infestations) | 8 | 10
Nausea (Gastrointestinal disorders) | 13 | 16
Diarrhea (Gastrointestinal disorders) | 10 | 11
Dizziness (Nervous system disorders) | 11 | 13
Fatigue (General disorders) | 9 | 10
Edema peripheral (General disorders) | 5 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.